CLINICAL TRIAL: NCT01022658
Title: Effects of Different Insulin Regimens on Artery Compliance, Endothelium Function and Autonomic Cardiac Function in Patients With Poorly Controlled Type 2 Diabetes: a Pilot Study
Brief Title: INSUlin Regimens and VASCular Functions
Acronym: INSUVASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P090303
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Type 2 Diabetes
Keywords: Insulin Therapy; Vago-sympathetic activity; arterial stiffness; endothelial function
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin; Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- detemir (Active Comparator): Insulin detemir at dinner or bedtime
  Interventions: Drug: Insulin
- aspart (Active Comparator): Insulin aspart before each meal
  Interventions: Drug: Insulin
- detemir and aspart (Active Comparator)
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — For diabetes treatment: metformin continued with insulin (according to arms)
  Other Names: LEVEMIR; NOVORAPID

SUMMARY:
Vago-sympathetic activity, arterial stiffness and endothelial function are integrators of cardiovascular risk. The aim of this pilot study is, in type 2 diabetic patients now requiring insulin, to compare the effects of improving glycemic control on these parameters with 3 different insulin regimens which will act especially at fasting or in post-prandial periods or both. Non invasive explorations will be performed before randomization and after 4 to 5 weeks of insulin therapy, at fasting and each hour after a standardized breakfast.

DETAILED DESCRIPTION:
Vago-sympathetic activity, arterial stiffness and endothelial function are integrators of cardiovascular risk. The effect of controlling fasting or post-prandial blood glucose or both on these parameters has not been studied in type 2 diabetic patients.

The aim of this pilot study is to compare the effects of improving fasting or post-prandial blood glucose glycemic control or both with 3 different insulin regimens for 4 to 5 weeks, on vago-sympathetic activity, arterial stiffness and endothelial function.

Patients will be recruited in the department of Endocrinology-Diabetology-Nutrition of Jean VERDIER hospital, AP-HP, and the department of Endocrinology and Metabolism of AVICENNE hospital, BOBIGNY, AP-HP, France. After an half day of cardiovascular explorations, 42 patients will be randomized in 3 groups determining their treatment for the following 4-5 weeks : insulin therapy with detemir at dinner or bed time, or with aspart at each meal, or with both of them.

Investigations will be performed in the morning 1) at the time of randomisation and 2) 4-5 weeks after the beginning of insulin therapy. We will evaluate at fasting and each hour after a standardized breakfast biological and metabolic parameters, arterial stiffness, endothelial function and nervous autonomic system with non-invasive devices: Sphygmocor®, Finapres®, laser-doppler et Endopat2000®. Body composition will be evaluated with impedance maestri and BodPod®.

ELIGIBILITY:
Inclusion Criteria:

* Consent patient
* Adults from 30 to 72 years old
* type 2 diabetic patients for at least 1 year
* able to self measure capillary blood glucose
* body mass index 20-37 kg/m²,
* HbA1c 7.1-12% under Metformin and SULFUNYREAS therapy for at least 2 months
* anti-hypertensive treatment or dyslipidemic treatment unchanged for 3 months

Exclusion criteria:

* pregnancy
* other antidiabetic medication in the previous 2 months,
* anti-hypertensive or lipid-lowering therapies having been changed in the previous 2 months,
* insulin allergy,
* uncontrolled preproliferative or proliferative diabetic retinopathy
* uncontrolled hypertension
* renal failure(creatinin clearance <40 ml/min)
* hepatocellular deficiency (prothrombin time <70%)
* anemia
* peripheral occlusive arterial disease
* cardiac arrhythmia

Ages: 30 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Vago-sympathetic activity, arterial stiffness, endothelial function | 4-5 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Valensi, Pr, Principal Investigator — CHU Jean VERDIER; Emmanuel Cosson, MD, PhD, Study Chair — CHU-Jean Verdier
Locations (1):
- Jean Verdier hospital, Department of Endocrinology-Diabetology-Nutrition, Bondy, France

REFERENCES:
- [Background] Nitenberg A, Cosson E, Pham I. Postprandial endothelial dysfunction: role of glucose, lipids and insulin. Diabetes Metab. 2006 Sep;32 Spec No2:2S28-33. doi: 10.1016/s1262-3636(06)70482-7. PMID 17375404
- [Background] Albertini JP, Valensi P, Lormeau B, Aurousseau MH, Ferriere F, Attali JR, Gattegno L. Elevated concentrations of soluble E-selectin and vascular cell adhesion molecule-1 in NIDDM. Effect of intensive insulin treatment. Diabetes Care. 1998 Jun;21(6):1008-13. doi: 10.2337/diacare.21.6.1008. PMID 9614623
- [Background] Valensi P, Cosson E. Hemodynamic changes in postprandial state. Diabetes Metab. 2006 Sep;32 Spec No2:2S37-41. doi: 10.1016/s1262-3636(06)70484-0. PMID 17375406
- [Background] Valensi P, Thi BN, Lormeau B, Paries J, Attali JR. Cardiac autonomic function in obese patients. Int J Obes Relat Metab Disord. 1995 Feb;19(2):113-8. PMID 7735337
- [Background] Dabire H, Brahimi M, Hadj-Brahim F, Le Clesiau H, Attali JR, Valensi P. [Role of vagosympathetic balance in obesity-induced hypertension]. Arch Mal Coeur Vaiss. 2004 Jul-Aug;97(7-8):749-52. French. PMID 15506059
- [Background] Valensi P, Paries J, Attali JR; French Group for Research and Study of Diabetic Neuropathy. Cardiac autonomic neuropathy in diabetic patients: influence of diabetes duration, obesity, and microangiopathic complications--the French multicenter study. Metabolism. 2003 Jul;52(7):815-20. doi: 10.1016/s0026-0495(03)00095-7. PMID 12870154
- [Background] Valensi P, Paries J, Lormeau B, Attia S, Attali JR. Influence of nutrients on cardiac autonomic function in nondiabetic overweight subjects. Metabolism. 2005 Oct;54(10):1290-6. doi: 10.1016/j.metabol.2005.04.016. PMID 16154426
- [Background] Ceriello A, Taboga C, Tonutti L, Quagliaro L, Piconi L, Bais B, Da Ros R, Motz E. Evidence for an independent and cumulative effect of postprandial hypertriglyceridemia and hyperglycemia on endothelial dysfunction and oxidative stress generation: effects of short- and long-term simvastatin treatment. Circulation. 2002 Sep 3;106(10):1211-8. doi: 10.1161/01.cir.0000027569.76671.a8. PMID 12208795
- [Background] Valensi P, Smagghue O, Paries J, Velayoudon P, Nguyen TN, Attali JR. Peripheral vasoconstrictor responses to sympathetic activation in diabetic patients: relationship with rheological disorders. Metabolism. 1997 Mar;46(3):235-41. doi: 10.1016/s0026-0495(97)90246-8. PMID 9054462
- [Background] Valensi P, Smagghue O, Paries J, Velayoudon P, Lormeau B, Attali JR. Impairment of skin vasoconstrictive response to sympathetic activation in obese patients: influence of rheological disorders. Metabolism. 2000 May;49(5):600-6. doi: 10.1016/s0026-0495(00)80034-7. PMID 10831169
- [Background] Sibony-Prat J, Paries J, Chabert M, Attali JR, Valensi P. [Alteration of cardiovascular vagosympathetic control evaluated by spectral analysis of variations of heart rate and blood pressure in obesity]. Arch Mal Coeur Vaiss. 1997 Aug;90(8):1155-8. French. PMID 9404427
- [Derived] Fysekidis M, Cosson E, Takbou K, Sutton A, Charnaux N, Banu I, Vicaut E, Valensi P. Effects of insulin analogs as an add-on to metformin on cutaneous microcirculation in type 2 diabetic patients. Microvasc Res. 2018 Mar;116:6-14. doi: 10.1016/j.mvr.2017.09.005. Epub 2017 Sep 24. PMID 28954218